CLINICAL TRIAL: NCT01983202
Title: Size at Birth in Newborn Children and Obstetric Outcomes in Women With PCOS
Brief Title: Obstetric Outcomes in Women With PCOS
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Marianne Andersen, Consultant, Odense University Hospital
Other Study IDs: 25624548
Record Dates: First submitted 2013-10-24; First posted 2013-11-13 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Polycystic Ovary Syndrome, PCOS
Keywords: PCOS; Pregnancy; Obstetric
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Women with PCOS: 208 women diagnosed with PCOS and giving birth after singleton pregnancies at Odense University Hospital during 2003-2011.
- Controls: 1040 women giving birth after singleton pregnancies at Odense University Hospital during 2003-2011, matched 1:5 to women with PCOS according to date-of-childbirth.

SUMMARY:
The aim of the study is to investigate body composition in newborn children of women with PCOS and controls and to investigate adverse obstetric outcomes in pregnant women with PCOS.

DETAILED DESCRIPTION:
A prospective cohort study investigating 208 women with PCOS giving birth after singleton pregnancies at Odense Univesity Hospital during 2003-2011 and a date-of-childbirth matched control group of 1040 women. Anthropometric data from children is recorded as well as data on maternal parity, age, pre-gestational BMI, and adverse obstetric outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with PCOS and giving birth during 2003-2011

Exclusion Criteria:

* Multiple pregnancy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 208 women diagnosed with PCOS at Department of Endocrinology and Metabolism and giving birth at Odense University Hospital during 2003-2011. Women with PCOS are matched 1:5 to a date-of-childbirth matched control group of 1040 pregnant women giving birth at Odense UNivesity Hospital.
Sampling Method: Probability Sample
Enrollment: 1248 (Actual)
Dates: Start 2003-01; Primary Completion 2011-01 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Anthropometric measures | Date of birth (1 day)
  Abdominal circumference, birth weight, birth length, and head circumference.

SECONDARY OUTCOMES:
Adverse obstetric outcomes | From beginning of pregnancy until the date of delivery (approximately 9 months)
  Presence of gestational diabetes mellitus, pregnancy induced hypertension, or pre-eclampsia during pregnancy. Registration of gestational age at childbirth, medical induction of birth, caesarean section,instrumental delivery, anal sphincter rupture, and shoulder dystocia.

OTHER OUTCOMES:
Neonatal complications | Date of birth (1 day)
  Registration of Apgar score 5 minutes after birth and admission to neonatal intensive care unit.

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Andersen, DMSci, Principal Investigator — Odense University Hospital
Locations (1):
- Department of Endocrinology, Odense University Hospital, Odense, Denmark